CLINICAL TRIAL: NCT00144248
Title: A Pharmacokinetic Study to Assess Nevirapine Levels in HIV-infected Patients With Impaired Hepatic Function
Brief Title: A Pharmacokinetic Study to Assess Nevirapine [Viramune] Levels in HIV Infected Patients With Impaired Hepatic Functions
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1100.1448
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: HIV Infections; Hepatic Insufficiency
MeSH Terms: conditions — HIV Infections; Hepatic Insufficiency | interventions — Nevirapine

INTERVENTIONS:
Drug: nevirapine

SUMMARY:
The objective of this study was to evaluate the steady-state clearance of nevirapine among HIV-1 positive patients with hepatic fibrosis, and to examine whether the degree of hepatic impairment influences clearance.

ELIGIBILITY:
INCLUSION

1. Male or female subjects >=18 years of age with HIV-1 infection and chronic liver disease as reflected by a documented biopsy with hepatic fibrosis present.
2. a. Participants must be receiving nevirapine 200 mg twice daily as part of a stable ARV regimen for a minimum of 6 weeks prior to trough level sample collection.

   b. Participants receiving nevirapine 400 mg once daily as part of a stable ARV regimen for a minimum of 6 weeks, who are willing to switch to nevirapi0 mg twice daily for a minimum of 14 days prior to trough collection.
3. Participants must have uoxylin and Eosin (H and E) stained slide and one trichrome stained pathology slide available at the time of enrollment. There is no time restriction on liver biopsy slides that pathologically confirm the presence of cirrhosis. The presence of cirrhosis must be documented on the liver biopsy report.

EXCLUSION

1. Current (within the past 4 weeks) HIV antiviral therapy with other NNRTI's.
2. Concurrent use (within the past 7 days) of any of the following:

   1. Systemic azole antifungal agents (fluconazole, itraconazole, ketoconazole, etc.)
   2. Clarithromycin
   3. Rifampin
   4. St John's Wort
3. Inability to provide a blood sample.
4. Patients who have evidence for hepatic or other encephalopathy above Grade 1
5. Patients with renal failure who require dialysis.
6. Pregnant and/or breast feeding women..

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2004-06-25 (Actual); Primary Completion 2006-06-01 (Actual)

PRIMARY OUTCOMES:
The primary endpoints are the degree of hepatic impairment, steady state nevirapine clearance, and the increase in estimated clearance when trough is supplemented by plasma levels measured one, two and four hours after nevirapine administration | Up to 4 hours

SECONDARY OUTCOMES:
Plasma levels of nevirapine metabolites of all patients and Child-Pugh scores among patients with cirrhosis. | Up to 14 hours

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — Boehringer Ingelheim
Locations (8):
- United States (5):
  - Boehringer Ingelheim Investigational Site, Bakersfield, California
  - Boehringer Ingelheim Investigational Site, San Francisco, California
  - California Pacific Medical Center, San Francisco, California
  - Albany Medical College, MC 142, Albany, New York
  - Boehringer Ingelheim Investigational Site, Providence, Rhode Island
- France (2):
  - Hopital de l'Hotel Dieu, Lyon
  - Hopital Pitie Salpetriere, Paris
- Hospital Clinico y Provincial de Barcelona - HIV, Barcelona, Spain

REFERENCES:
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/19620337